CLINICAL TRIAL: NCT06417242
Title: Predicting Outcomes in Atrial Fibrillation and Heart Failure
Acronym: PrOAF-HF
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 318987
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: ablation; atrial fibrillation; AF; heart failure; HF; rhythm control
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF index disease: Patients with no history of atrial fibrillation at the time of first diagnosis of heart failure
- Unclear index disease: Patients in whom the index disease is unknown or in whom atrial fibrillation is the index disease

SUMMARY:
PrOAF-HF will aim to test if rhythm control delivered through catheter ablation in patients in whom it is not clear whether atrial fibrillation or heart failure were the first disease results in a greater improvement in left ventricular ejection fraction (LVEF) compared with patients where heart failure was diagnosed first with no evidence of AF.

DETAILED DESCRIPTION:
Heart failure is a chronic disease affecting half a million patients in the UK. Up to 40% of patients with heart failure also suffer from atrial fibrillation. A subgroup of patients with atrial fibrillation and heart failure have tachycardia induced cardiomyopathy and benefit from significant improvement of the left ventricular function with restoration of sinus rhythm. Currently those patients can only be identified based on their response to treatment. Investigators aim to improve the treatment of AF-HF patients. The group will develop a robust modelling framework for simulating the hearts of AF-HF patients' hearts to predict patients' response to therapy and infer patient history. This modelling framework will enable integration of predictive simulations into clinical study design where the inferred initiating disease and predicted patient response to therapy are tested for selecting either rate or rhythm control in AF-HF patients.

The primary objective is to test if rhythm control delivered through catheter ablation in patients where either the index disease is unclear or where AF was diagnosed prior to the onset of HF improves LVEF more than in patients where HF was diagnosed first with no evidence of AF.

The secondary objectives are to examine whether the ability to terminate AF during pulmonary vein isolation is influenced by the identified index disease and to determine whether the identified index disease affects AF recurrence rate at 6 months and/or burden post ablation. This study will also identify whether the index disease affects pressure measurements as predictors of change in ejection fraction, hospitalisation, and death rates during the follow up period.

This will be a non-interventional cohort study. Routinely acquired clinical data collected during pre-procedure work up will be accessed for research purposes including: 24-48 hour ambulatory (Holter) monitoring, electrocardiograph (ECG) in AF and in sinus rhythm if available; echocardiography, and clinical history and examination details.

Additionally, an atrial cardiac magnetic resonance imaging (MRI) scan will be performed including assessment of atrial structure, function, fibrosis and epicardial fat burden. Symptom questionnaires will be performed During the ablation procedure, additional time will be taken to perform electrophysiological assessment in all four chambers of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent AF
* LVEF ≤40% prior to commencement of treatment
* NYHA class ≥2
* Patient must have been commenced on guideline directed medical therapy (GDMT)
* Patient planning to proceed to radiofrequency atrial fibrillation ablation
* Age 18-80 years
* Able and willing to provide written informed consent

Exclusion Criteria:

* Any clinical contra-indication to ablation
* Any disease limiting life expectancy to <1 year
* Potential participant currently pregnant or breast feeding
* Contraindication to MRI
* Paroxysmal or permanent AF
* Unable to understand verbal or written explanations given in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosis of both heart failure and atrial fibrillation, listed for atrial fibrillation ablation will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in LVEF | 6 months post ablation
  Change in left ventricular ejection fraction measured on echocardiography

SECONDARY OUTCOMES:
Immediate change in LVEF | Immediately post procedure
  Change in left ventricular ejection fraction on echocardiography
AF recurrence | 6 months post ablation
  Presence of AF
Termination of AF during the procedure | Intraprocedural
  Termination of AF during the ablation procedure
Hospitalization | 6 months
  Hospitalization for any reason
Death | 6 months
  Death of any cause and cardiovascular death
Pressure measurements as predictors of change in LVEF | Intraprocedural measurements - change in LVEF as above
  Invasive measurements of all four chambers pressure changes during the ablation
Change in atrial fibrillation burden | 6 months post ablation
  Change in atrial fibrillation burden assessed on a continuous Holter monitor
Change in symptoms | 6 months post ablation
  Change in quality of lide questionnaire scores